CLINICAL TRIAL: NCT06167512
Title: Metabolic Reprogramming in Renal Tubular Cells in Acute Kidney Injury Following Severe Trauma
Acronym: METAKIT
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231084; 2023-A01597-38 (Other: IDRCB)
Record Dates: First submitted 2023-11-21; First posted 2023-12-12 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Multi-organ Failure After Severe Trauma
Keywords: Severe trauma; hemorrhagic shock; Acute kidney Injury; Acute respiratory distress syndrome; Multi-organ failure
MeSH Terms: conditions — Wounds and Injuries; Shock, Hemorrhagic; Acute Kidney Injury; Respiratory Distress Syndrome; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- polytrauma patients: polytrauma patients
- healthy volunteers: healthy volunteers

SUMMARY:
Severe trauma remains the leading cause of death in people under 50, and is associated with high morbidity, including severe disability, with a substantial socio-economic impact. Secondary to trauma, multiple mechanisms (inflammatory, ischemic, oxidative, etc.) setting in rapidly, leads to organ failure, one of the three first cause of death. Vascular damage, with vasoplegia, renal damage, with acute kidney injury (AKI), and pulmonary damage, with acute respiratory distress syndrome (ARDS), are the most frequently observed but all organs can be affected whatever the type of trauma. For these reasons, identifying the pathophysiological pathways involved in organ failure induced by severe trauma is a major step towards limiting the morbidity and mortality induced by trauma, and proposing therapies to prevent them.

Because of the variability of lesions in these patients, and the multiplicity of pathways activated, the mechanisms involved and their causality with organ failure following severe trauma, are still poorly understood. Given their frequency and importance in terms of morbidity and mortality, the investigators decided to take a particular interest in the mechanisms leading to renal and pulmonary injury. The investigators' hypothesis is that the study of urinary and blood markers not performed as part of clinical routine would provide a better understanding of the pathophysiological mechanisms leading to organ failure secondary to severe trauma, and more specifically to renal and pulmonary injuries. With TRAUMATEC study, the investigators will explore mechanisms leading to AKI and ARDS through blood and urine samples of 60 severe trauma patients sampled over the first 48 hours after ICU admission and a reference of 20 healthy volunteers.

DETAILED DESCRIPTION:
The investigators plan to include 60 patients over 18 years old with severe trauma, defined with an ISS≥9 and 20 healthy volunteers 18 years old as a reference group.

Blood and urine samples will be collected at ICU arrival, 12-, 24- and 48- hours after ICU admission. Specific dosages will then be realized on blood and urines to study metabolic and hormonal pathway leading to AKI and ARDS.

The primary objective of the study is to explore the association between renal metabolic changes and renal function impairment following severe trauma.

Secondary objectives are (1) to explore mitochondrial changes observed at the renal cellular level, on in vitro renal culture cells after exposure to trauma patient serum (2) to explore the association between plasma metabolic changes and renal and pulmonary function impairment following severe trauma (3) to explore the association between hormonal metabolic changes and renal and pulmonary function impairment following severe trauma (4) to explore the association between red blood cell-induced oxidative stress and renal function impairment following severe trauma (5) to explore the association between changes in the hemoglobin recycling (chelation) system and impaired renal function following severe trauma (6) to explore renal tubular damage secondary to severe trauma (7) to explore the pathophysiological mechanisms associated with pulmonary damage following severe trauma (8) to describe mortality at day 30.

ELIGIBILITY:
Inclusion Criteria:

Trauma patients :

* Adult patients (age ≥ 18 years)
* Patient admitted for suspected severe trauma (1 Vittel criteria)
* Injury Severity Score ≥ 9
* Health insurance
* Written consent obtained from the patient or trusted support person / family member / close friend, or inclusion in an emergency situation and written consent obtained from the patient (trusted support person / family member / close friend if necessary) as soon as possible (article L1122-1-2 of the CSP).

Healthy volunteers :

* Adult patients (≥ 18 years)
* Affiliated with health insurance
* Written informed consent́
* Patient respecting matching

Exclusion Criteria:

Trauma patients :

* Pregnant patient
* Minor patient
* Adult under guardianship, curatorship or safeguard of justice
* Patient under Aide Médicale d'État
* Chronic renal failure on dialysis
* Chronic respiratory disease
* Patient with chronic cardiac insufficiency
* Systemic inflammatory disease

Healthy volunteers :

* Pregnant patient
* Minor patient
* Adult under guardianship, curatorship or safeguard of justice
* Patient under Aide Médicale d'État
* Patient with chronic renal failure on dialysis
* Chronic respiratory disease
* Patient with chronic cardiac insufficiency
* Systemic inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: polytrauma patients : a population of severe trauma patients at risk of failure secondary organs.
  healthy volonteers
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-09-27 (Estimated); Study Completion 2025-10-27 (Estimated)

PRIMARY OUTCOMES:
Profile of urinary metabolite concentrations measured by mass spectometry | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Metabolomic study of patients urine according to AKI and compared to healthy volunteers measured by mass spectometry

SECONDARY OUTCOMES:
mitochondrial enzymatic activities of cultured Human Kidney 2 (HK2) kidney cells exposed to patient serum and exposed to serum from healthy volunteers | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  In vitro mitochondrial function of cultured Human Kidney 2 (HK2) kidney cells exposed to patient serum and exposed to healthy volunteer serum assessed by enzymatic activities by Seahorse XFe96 analyzer
mitochondrial membrane potential of cultured Human Kidney 2 (HK2) kidney cells exposed to patient serum and exposed to serum from healthy volunteers | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  In vitro mitochondrial function of cultured Human Kidney 2 (HK2) kidney cells exposed to patient serum and exposed to healthy volunteer serum assessed by measurement of mitochondrial membrane potential by fluorescence
mitochondrial Adenosine TriPhosphate (ATP) content of cultured Human Kidney 2 (HK2) kidney cells exposed to patient serum and exposed to serum from healthy volunteers | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  In vitro mitochondrial function of cultured Human Kidney 2 (HK2) kidney cells exposed to patient serum and exposed to healthy volunteer serum assessed by measurement of ATP content by spectrofluorimetry
expression levels of mitochondrial of cultured Human Kidney 2 (HK2) kidney cells exposed to patient serum and exposed to serum from healthy volunteers | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  In vitro mitochondrial function of cultured Human Kidney 2 (HK2) kidney cells exposed to patient serum and exposed to healthy volunteer serum assessed by measurement of expression levels of mitochondrial by Western-blot
Plasma metabolite concentration profile measured by mass spectrometry | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Metabolomic study of patients plasma measured by mass spectrometry according to AKI and ARDS and compared to healthy volunteers
advanced glycation end products (AGEs) produced by red blood cells | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Measurement of oxidative stress produced by red blood cells assessed by advanced glycation end products (AGEs)
reactive oxygen derivatives produced by red blood cells | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Measurement of oxidative stress produced by red blood cells assessed by reactive oxygen derivatives
erythrocyte NO production produced by red blood cells | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Measurement of oxidative stress produced by red blood cells assessed by erythrocyte NO production
haptoglobin level | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Hemoglobin recycling system assessed by haptoglobin
haptoglobin-hemoglobin complexes level | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Hemoglobin recycling system assessed by haptoglobin-hemoglobin complexes
free hemoglobin level | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Hemoglobin recycling system assessed by free hemoglobin
monocyte CD163 receptor from peripheral blood mononuclear cell (PBMC) isolation level | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Hemoglobin recycling system assessed by monocyte CD163 receptor from peripheral blood mononuclear cell (PBMC) isolation
Heme oxygenase-1 (HO-1) enzyme catabolizing heme level | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Hemoglobin recycling system assessed by Heme oxygenase-1 (HO-1) enzyme catabolizing heme
renin-angiotensin-aldosterone (RASS) profile | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Measurement of RASS
Antidiuretic hormone (ADH) profile | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Measurement of ADH
cortisol profile | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Measurement of cortisol
leptine profile | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Measurement of leptine
Intensity of renal tubular injury | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Renal tubular injury assessed by standard urinary markers: neutrophil gelatinase-associated lipocalin (NGAL), Kidney injury molecule 1 (KIM-1), IGFB-7, tissue inhibitor of metalloproteinases-2 (TIMP-2), cystatin C
hypoxemia level | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Pulmonary injury during hospitalization in intensive care evaluated by hypoxemia assessed by the PaO2/FiO2 ratio
use of mechanical ventilation | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Pulmonary injury during hospitalization in intensive care evaluated by use of mechanical ventilation
Radiographic Assessment of Lung Edema (RALE) score | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Pulmonary injury during hospitalization in intensive care evaluated by Radiographic Assessment of Lung Edema (RALE) score
alveolar epithelial lesions | On admission, at 12 hours, 24 hours and 48 hours of hospital admission
  Pulmonary injury during hospitalization in intensive care evaluated by evaluation of alveolar epithelial lesions by circulating soluble Receptor for Advanced Glycation Endproducts (sRAGE) assay.
Death | Day 30
  Vital status at day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Bicetre hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Undecided